CLINICAL TRIAL: NCT06297980
Title: Impact of MEnstruation on Glycemic Response and Exercise In Females With Type 1 Diabetes
Acronym: MERIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-1513
Record Dates: First submitted 2024-02-12; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Type 1 Diabetes; Hypoglycemia; Hyperglycaemia Due to Type 1 Diabetes Mellitus; Menstruation Disturbances
Keywords: type 1 diabetes; menstrual cycle; exercise; hypoglycemia; hyperglycemia; glucose control
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Menstruation Disturbances; Motor Activity; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: This will be a parallel group randomized control trial of a personalized glucose control intervention to target changes in glycemic control related to the menstrual cycle that are identified during a 3 month observational period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized treatment (Experimental): We will test an intervention that includes up to four personalized adjustments to food intake, insulin dose and glycemic algorithms by menstrual cycle phase, based on the three months of observational data collected.
  Interventions: Other: Personalized modifications to treatment to address menstrual cycle effects on glycemia
- Standard Care (No Intervention): In this arm, women will continue with their usual insulin dose, food intake and glycemic algorithms as determined by their provider

INTERVENTIONS:
Other: Personalized modifications to treatment to address menstrual cycle effects on glycemia — The study physician will examine glucose patterns measured using continuous glucose monitoring over a 3 month observational period to identify hypo- or hyperglycemia related to menstrual cycle phase or exercise, and will provide changes to insulin basal or bolus rates, carbohydrate ratios, post-exercise food intake or use of sleep mode on automated insulin delivery systems.
  Arms: Personalized treatment

SUMMARY:
The objectives of this study are to examine how sex hormones (use of hormonal birth control, menstrual cycle phase) impact glycemic control among women with type 1 diabetes (T1D), and to test adjustments to insulin dosing and food intake to ameliorate cycle-related glycemic variability. A secondary aim is to examine how the menstrual cycle and use of hormonal birth control impact patient-reported outcomes and glycemic responses to physical activity.

DETAILED DESCRIPTION:
The overall goal of this project is to further understand the impact of hormonal status on glycemic metrics and to test personalized changes to insulin dosing, through implementing the following specific aims:

Specific Aim 1: Using CGM, examine glucose levels among women with T1D by menstrual cycle phase over a three month period to establish baseline glycemic variability, to identify personalized patterns of glycemic control across the menstrual cycle phase, and to test glycemic responses to acute bouts of aerobic, interval and resistance training.

Specific Aim 2: Using the data from the observational period, examine patterns of glycemic variability by menstrual cycle phase in order to determine the appropriate alteration to insulin delivery needed to improve glycemic control across the menstrual cycle among women with T1D

Specific Aim 3: Test an intervention that includes up to four personalized adjustments to food intake, insulin dose and glycemic algorithms by menstrual cycle phase in a randomized intervention and control group. We will also examine responses to daily activity, planned exercise activities, and acute bouts of aerobic, interval and resistance exercise.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-45 who have had type 1 diabetes for at least 12 months
* Premenopausal with either menstrual cycles or currently using oral contraceptives

Exclusion Criteria:

* Women who are postmenopausal, pregnant, trying to become pregnant, or have had a hysterectomy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Glucose time in range | 3 months during randomization to intervention or standard care
  time spent with glucose 70-180mg/dL on continuous glucose monitor
Glucose standard deviation | 3 months during randomization to intervention or standard care
  standard deviation (mg/dL) of glucose on continuous glucose monitor

SECONDARY OUTCOMES:
Mean glucose (mg/dL) pre-exercise | mean glucosewithin 5 minutes of beginning planned exercise bouts based on start time reported by study participant and/or accelerometer data
  Mean glucose from continuous glucose monitor in response to exercise
Mean glucose (mg/dL) while exercising | mean glucose measured every 5 minutes while actively exercising (between exercise start and end times as reported by study participant or based on accelerometer data, from a minimum of 5 minutes to up to 480 minutes)
  Mean glucose from continuous glucose monitor in response to exercise
Mean glucose (mg/dL) over 24 hours after exercise | mean glucose during the 24 hours after beginning planned exercise bouts (from participant reported or acceleromater data based start of exercise to 24 hours later)
  Mean glucose from continuous glucose monitor in response to exercise
Glucose standard deviation | glucose standard deviation during the follicular (starting day one of the menstrual period as self-reported by study participant through a positive home test for ovulation by participant, or for a maximum of 30 days if no positive ovulation test)
  standard deviation (mg/dL) of glucose on continuous glucose monitor
Glucose standard deviation | glucose standard deviation during the luteal menstrual cycle phase (starting from the day of a positive home ovulation test to the start of the next period reported by participant, for a maximum of 30 days if no next period begins)
  standard deviation (mg/dL) of glucose on continuous glucose monitor

CONTACTS AND LOCATIONS:
Overall Officials: JANET K SNELL-BERGEON, PhD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
There will be a steering committee that will review requests for individual participant data through an ancillary study and paper proposal process
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will become available within 12 months from the end of the data collection
Access Criteria: Researchers wishing to access IPD will be requested to complete an application and a data transfer agreement